CLINICAL TRIAL: NCT04019951
Title: The Effect of a Standardized Liquid Breakfast Containing a Propionate Colon Release Form on ad Libitum Eating and Appetite Perception in Healthy Overweight Humans: A Double-blinded, Randomized, Cross-over Study.
Brief Title: The Effect of a Propionate Colon Release Form on ad Libitum Eating and Appetite Perception
Acronym: METABIOTIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2016-11-28-PROP
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propionate (1 g) (Experimental): Participants will receive 1 g of Ca-propionate in a colon-release form. Volunteers will receive the product on visits 2, 3 and 4. Each of the visits will be separated by > 5 days. Visit 5, the end of study visit, will occur within 5 days of visit 4.
  Interventions: Dietary Supplement: Ca-propionate 1 g
- Propionate (3 g) (Experimental): Participants will receive 3 g of Ca-propionate in a colon-release form. Volunteers will receive the product on visits 2, 3 and 4. Each of the visits will be separated by > 5 days. Visit 5, the end of study visit, will occur within 5 days of visit 4.
  Interventions: Dietary Supplement: Ca-propionate 3 g
- Placebo (Placebo Comparator): Participants will receive 2.6 g of cellulose in a colon-release form. Volunteers will receive the product on visits 2, 3 and 4. Each of the visits will be separated by > 5 days. Visit 5, the end of study visit, will occur within 5 days of visit 4.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ca-propionate 1 g — 1 g of Ca-propionate will be mixed in 203 mL of a standardized liquid breakfast
  Arms: Propionate (1 g)
Dietary Supplement: Ca-propionate 3 g — 3 g of Ca-propionate will be mixed in 203 mL of a standardized liquid breakfast
  Arms: Propionate (3 g)
Dietary Supplement: Placebo — 2.6 g of cellulose will be mixed in 203 mL of a standardized liquid breakfast
  Arms: Placebo

SUMMARY:
The present study aims to investigate the effect of a standardized liquid breakfast containing a food grade propionate colon release form on ad libitum eating and appetite perception in healthy overweight humans using a double-blinded, randomized, cross-over study design

DETAILED DESCRIPTION:
To determine, in healthy overweight subjects, the acute effect of a standardized liquid breakfast containing a propionate colon release form compared with placebo on appetite and GI comfort, food intake, serum glucose and insulin, plasma ghrelin, total GLP-1 and serum PYY concentrations, and plasma propionate concentrations

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females, 18-60 years of age
2. Body mass index (BMI) ≥25 and <30 kg/m² at screening.
3. Unrestrained eater (Score of ≤11 on the Eating Habits Questionnaire)
4. Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
5. Subject is willing to abstain from strenuous exercise, and consume alcoholic drinks 24 hours before study days and during study days.
6. Willing to refrain from dietary supplement that are known to affect appetite (e.g. some herbal supplements), from prebiotic and probiotic supplements and large amounts of dietary fiber (inulin, metamucil, oat bran, etc) throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
7. Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
8. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.
9. Subject regularly has at least one bowel movement per day

Exclusion Criteria:

1. Smokers
2. Haemoglobin measurements of <120g/L for females and <130g/L for males (as per WHO criteria for anaemia).
3. Fasting serum glucose (above or equal to 7.0mmol/L). AST, ALT, GGT and ALP >1.8 times upper limit of normal; creatinine >1.2 times upper limit of normal; fasting triglycerides >4.0 mmol/L; and electrolytes outside the normal range.
4. Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
5. Use of medications/dietary supplements known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might: 1) make participation dangerous to the subject or to others, or 2) affect the results as judged by the Investigator.
6. History of propionic acidemia.
7. Major trauma or surgical event within 3 months of screening.
8. Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
9. Known intolerance, sensitivity or allergy to any ingredients in the study products.
10. Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc).
11. Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg as defined by the average blood pressure measured at screening.
12. Change in body weight of >3.5kg within 4 weeks of the screening visit.
13. Presence of any signs or symptoms of an active infection within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment (i.e. antibiotic therapy) has been completed at least 4 weeks prior to each test visit.
14. History of cancer in the prior two years, except for non-melanoma skin cancer.
15. Recent history (within 12 months of screening) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as > 14 drinks per week (1 drink=12 oz beer, 5 oz wine, or 1.5 oz distilled spirits).
16. Exposure to any non-registered drug product within 30 d prior to screening.
17. Subject has donated more than 300 mL of blood during the three months prior to screening.
18. Any history of an eating disorder (eg. anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a health professional

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Ad-libitum energy intake | t=210 minutes
  Ad-libitum energy intake will be assessed by giving subjects a choice of an excess of individual pizza slices

SECONDARY OUTCOMES:
Subjective ratings of appetite and GI comfort | Every 30 minutes during an interval of 6 hours
  Subjective measurements of motivation to eat and GI physical comfort will be assessed using validated questionnaires, i.e. Visual Analog Scales (VAS). Each of the questions on the VAS is a 100 mm line anchored at each end with opposing statements. Participants mark a vertical line on the line at a point that they felt reflect their feelings at the moment the test was taken. Scores will be assessed by measuring the distance between the intersection of the vertical line with the line and the left end of the line. VAS include a set of questions, such as feelings of fullness, feelings of hunger, prospective food consumption.
24 h food intake | Food intake is recorded from the time of the start of the ad-libitum food test until 24 hours later
  Completion of a food diary
Serum glucose | Every 30 minutes during an interval of 6 hours
  Serum glucose analysis will be done using either the Vitros 350 Chemistry System or an YSI model 2300/2700 STAT analyser
Plasma insulin | Every 30 minutes during an interval of 6 hours
  Plasma insulin will be measured using an insulin ELISA Immunoassay kit
Plasma ghrelin | Every 30 minutes during an interval of 6 hours
  Immunoassay kits will be used to measure plasma ghrelin
Plasma total glucagon-like peptide-1 (GLP-1) | Every 30 minutes during an interval of 6 hours
  Immunoassay kits will be used for measure plasma total GLP-1
Plasma peptide YY (PYY) | Every 30 minutes during an interval of 6 hours
  Immunoassay kits will be used for measure plasma PYY
Plasma propionate | Every 30 minutes during an interval of 6 hours
  Plasma propionate will be measured using HPLC MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, Principal Investigator — GI Labs
Locations (1):
- GI Labs, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No